CLINICAL TRIAL: NCT03012659
Title: Contraceptive Equity Study
Brief Title: Contraceptive Equity Study 2016
Acronym: CES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Planned Parenthood Federation of America (Other)
Collaborators: Planned Parenthood South Atlantic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00019792
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Contraception Behavior; Contraceptive Usage; Contraceptive Method Switching
Keywords: contraceptive counseling; cluster randomized trial; provider counseling training
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Full-day contraceptive counseling training for health center staff
  Interventions: Behavioral: Contraceptive Counseling Training
- Control Arm (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Contraceptive Counseling Training — Intervention sites will receive:
  1. In person training: All staff at an intervention health center will participate in a one-day counseling training.
  2. On-site shadowing: Trainers will shadow staff in-clinic the day following the training to observe the counseling implementation and provide additional coaching and support.
  3. Technical assistance: A Planned Parenthood clinic operations expert will provide follow-up technical assistance.
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to assess the impact of a provider counseling training on patient contraceptive behaviors and satisfaction in a clustered randomized trial among 10 Planned Parenthood health centers.

DETAILED DESCRIPTION:
This study builds upon prior research on a contraceptive counseling protocol and training developed and studied by partners at New York University and Planned Parenthood Federation of America. This contraceptive counseling protocol is informed by the literature on contraceptive behavior, expertise in decision and communication science, and formative qualitative research with Planned Parenthood providers and patients. Jaccard et al. (in press) conducted a cluster randomized control study of the counseling intervention with 10 Planned Parenthood health centers, where staff at intervention sites participated in a one-day training on the counseling protocol followed by a day of in-clinic shadowing. Patients were enrolled on-site and contacted for follow-up at six months and 12 months.

Results of this study indicated that patients at intervention sites were more satisfied with their contraceptive counseling and method choice, and at one or both follow-ups there were fewer gaps in contraceptive protection, more dual method use, and less non-use of birth control. There was no significant difference in accurate use of birth control pills.

Planned Parenthood Federation of America (PPFA) adapted and piloted training in this contraceptive counseling protocol during 2016 with 18 Planned Parenthood affiliated organizations across the country. This training was integrated into a one-day event that also included a provider training to address barriers in access to intrauterine devices and implants. A mixed-methods implementation evaluation was conducted to assess outcomes for staff and patients and identify challenges in implementation. Preliminary findings from the program pilot year demonstrated positive trends for outcome measures, produced lessons learned on implementation challenges, and provided support for new adaptations to the training program and counseling protocol. The previous pilot year evaluation was designed to assess patient satisfaction and method choice before and after the training, but could not answer questions about continued impact on other outcomes of interest. The current study will use a cluster randomized control design with 10 Planned Parenthood health centers to assess patient outcomes. Five health centers randomized to the intervention will receive the contraceptive counseling training. As the control group, the other five health centers will conduct usual care. Women will be enrolled onsite at the health center and then contacted for follow-up at approximately 30 and 90 days post-enrollment. Target enrollment is 100 women per site (1000 total).

ELIGIBILITY:
Inclusion Criteria:

* Females who have received contraceptive counseling at participating health centers.
* Ability to understand written and spoken English.

Exclusion Criteria:

* Non-English speakers

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Contraceptive Continuation | 3 months
  Patient-reported contraceptive continuation

SECONDARY OUTCOMES:
Method Satisfaction | 1 month and 3 months
  Patient-reported satisfaction with contraceptive method
Dual-Use | 1 month and 3 months
  Patient-reported dual-use of condoms plus other method
Missed Pills | 1 month and 3 months
  Number of patient-reported missed oral contraceptive pills among pill users
Method Switching | 1 month and 3 months
  Patient-reported method switching
Patient experience of counseling best practices during their visit | Baseline
  Patient-report of staff implementation of the best counseling practices during their visit

OTHER OUTCOMES:
Access to same-day services for all contraceptive methods | Baseline
  Patient report of being offered to start method on same day as their visit (if desired)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah R. Simons, DrPH, Principal Investigator — Planned Parenthood Federation of America
Locations (1):
- Planned Parenthood South Atlantic, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No